CLINICAL TRIAL: NCT06110923
Title: A Randomized, Open-label and Parallel Study to Evaluate the Pharmacokinetics and Safety of CKD-846 in Healthy Male Subjects
Brief Title: A Clinical Trial to Compare and Evaluate Evaluate the Pharmacokinetics and Safety of CKD-846
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A133_01PK2306
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostate Hypertrophy(BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A1 (Test group) (Experimental): CKD-846 A, Single dose
  Interventions: Drug: CKD-846
- R (Reference group) (Experimental): D091, Multi dose
  Interventions: Drug: D091
- A2 (Test group) (Experimental): CKD-846 A, Single dose
  Interventions: Drug: CKD-846
- B2 (Test group) (Experimental): CKD-846 B, Single dose
  Interventions: Drug: CKD-846
- A3 or B3 (Test group) (Experimental): CKD-846 A or B, Single dose
  Interventions: Drug: CKD-846

INTERVENTIONS:
Drug: CKD-846 — once administration of Investigational Product
  Other Names: Investigational Product(Test)
  Arms: A1 (Test group); A2 (Test group); A3 or B3 (Test group); B2 (Test group)
Drug: D091 — once administration of Investigational Product per day
  Other Names: Investigational Product(Reference)
  Arms: R (Reference group)

SUMMARY:
A Clinical trial to compare and evaluate evaluate the pharmacokinetics and safety of CKD-846

DETAILED DESCRIPTION:
A randomized, open-label and parallel study to evaluate the pharmacokinetics and safety of CKD-846 in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man aged between 19 to 55 at screening
2. Weight ≥ 55kg
3. Body mass index (BMI) of 18.5 to 27.0kg/m2
4. Those who agree to contraception from the first Investigational Product (IP) dosing day till 6 months after the last dosing day and decide not to provide sperm during the participation of clinical trial
5. Those who voluntarily decide to participate in paper and agree to comply with the cautions after fully understand the detailed description of this clinical trial

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of Hepatopathy, Renal, Neurological, Immunity, Respiratory, Endocrine, urinary, tumor or Psychical disorder
2. Those who have a history of clinically significant cardiovascular diseases such as myocardial infarction, angina pectoris, ventricular arrhythmia, heart failure, left ventricular outflow tract stenosis, stroke, and transient ischemic attack within 2 years prior to the first administration of the investigational drug

   * Those who have had myocardial infarction within the last 90 days
   * Those who have had unstable angina or angina that occurred during sexual intercourse
   * Those who have had heart failure of New York Heart Association class 2 or higher in the past 6 months
   * Those who have had a stroke within the last 6 months
3. Those with the following eye diseases

   * Those with known genetic degenerative retinal diseases, including retinitis pigmentosa
   * People who have lost vision in one eye due to non-arteritic anterior ischemic optic neuropathy
4. Those with a past history of erection lasting more than 4 hours and priapism (erection accompanied by pain for more than 6 hours) while taking PDE5 inhibitors such as tadalafil
5. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery which can interfere with drug absorption
6. Persons with a history of clinically significant hypersensitivity to drugs or additives, including ingredients of clinical investigational drugs
7. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
8. A person who is judged to be unsuitable as a test subject in a screening test (screening items such as questionnaire, blood pressure, 12-lead ECG, physical examination, clinical laboratory test, etc.) conducted within 28 days before administration of the investigational drug

   * Aspartate aminotransferase (AST), Alanine aminotransferase (ALT) > 1.5 times higher than upper normal level
   * Total bilirubin > 1.5 times higher than upper normal level
   * Epidermal Growth Factor Receptor (eGFR) (estimated Glomerular Filtration Rate, which is calculated by MDRD) < 60 mL/min/1.73m2
   * "Positive" or "Reactive" test result of Hepatitis B & C, HIV, rapid plasma reagin test (RPR) > 10.0 ng/mL
   * Prostate specific antigen (PSA)
   * Under 5 min resting condition, systolic blood pressure >150 mmHg or or <90 mmHg, diastolic blood pressure >100 mmHg or <50mmHg.
9. Those who has a drug abuse history within one year or positive reaction on urine drug screening test.
10. Those who have taken the following drugs, excluding topical drugs without significant systemic absorption, within the relevant period and it is judged that the administered drugs may affect this study or affect the safety of subjects

    * Over the counter (OTC), vitamins, health supplement within 7 days before the first dose of the investigational drug
    * Ethical drug (ETC), herbal medicinal preparations within 14 days before the first dose of the investigational drug
    * CYP3A4 inhibitors or CYP3A4 inducers within 30 days before the first dose of the investigational drug
    * Depot injection or implantation within 30 days before the first dose of the investigational drug
11. Persons who must take the following drugs regularly and/or intermittently during the clinical trial period

    * Nitrate preparations or NO donors
    * Alpha blockers
    * GC stimulators
12. Those who continuously smoke excessively or consume caffeine or alcohol (cigarettes: >10 cigarettes/day, caffeine: >5 cups/day, alcohol: >210 g/week)
13. A person who consumed food containing grapefruit within 7 days before the first administration of the investigational drug (e.g., a person who consumed more than 1L of grapefruit-containing beverages per day within 7 days before the first administration of the investigational drug)
14. Persons who participated in another clinical trial (including bioequivalence test) and received an investigational drug within 180 days prior to the date of first administration of the investigational drug (in the case of biological products, the period may be extended considering the half-life)
15. Those who donated whole blood within 60 days before the first date of administration and donated ingredients within 30 days
16. Those who have received blood transfusion in 30 days
17. Those who are deemed insufficient to participate in clinical study by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 31 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of CKD-846 | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Concentration of During the administration period
Concentration of D091 | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Concentration of During the administration period

SECONDARY OUTCOMES:
CKD-846 of AUCinf | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Area under the curve
CKD-846 of Tmax | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Time to maximum plasma concentration
CKD-846 of t1/2 | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Terminal elimination half-life
CKD-846 of CL/F | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Apparent clearance of drug in plasma
CKD-846 of Vd/F | Pre-dose, Post-dose 0.33, 0.67, 1, 1.5, 2, 3, 4, 6, 10, 24 hours (During the administration period)
  Apparent volume of distribution
D091 of Cmax | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Maximum concentration of drug in plasma
D091 of AUCt | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Area under the curve
D091 of AUCinf | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Area under the curve
D091 of Tmax | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Time to maximum plasma concentration at steady state
D091 of t1/2 | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Terminal elimination half-life
D091 of CL/F | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Apparent clearance of drug in plasma
D091 of Vd/F | Pre-dose, Post-dose 0.5, 1, 2, 4, 6, 10, 24, 48, 72, 96 hours (During the administration period)
  Apparent volume of distribution

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No